CLINICAL TRIAL: NCT03709862
Title: Whole Genome Sequencing of Syphilis Using Routine Clinical Samples
Brief Title: Global Syphilis Sequencing
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 16014
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Residual DNA from routine clinical samples (lesion swabs/serum) of patients with Syphilis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Syphilis: Patients with syphilis and detectable Treponema pallidum DNA in a routinely collected clinical sample
  Interventions: Diagnostic Test: Whole Genome Sequencing

INTERVENTIONS:
Diagnostic Test: Whole Genome Sequencing — Residual DNA from clinical samples will be utilised for whole genome sequencing of Treponema pallidum the causative agent of syphilis

SUMMARY:
Syphilis is an important sexually transmitted infection. There has been an epidemic of syphilis amongst men who have sex with men in the United Kingdom in the last decade. Early infection with syphilis causes a genital ulcer followed, in the absence of treatment, by a generalised illness often accompanied by rash. Studies on syphilis have been limited because it is not possible to grow syphilis outside of the body. New approaches allow the whole genetic sequence of Treponema pallidum to be obtained from a swab.

In this study residual DNA collected as part of routine patient care of patients seen at sexual health clinics in the UK will be used for sequencing. No patient contact is involved in the study which is limited to whole genome sequencing using residual material from samples. By better understanding the genome of the T.pallidum insights will be gained in to the pathogenesis of this important sexually transmitted disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of syphilis

Exclusion Criteria:

* No PCR positive clinical sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to sexual health services in UK with a diagnosis of syphilis.
  We will identify residual T.pallidum DNA from routinely collected clinical samples held at participating clinics/hospitals. Data accompanying these samples will be anonymised and will not include patient identifiable information. Accompanying data will include: city of origin, age, gender, HIV status and sexual orientation.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Genomic Diversity of Treponema Pallidum as assessed by nucleotide diversity and phylogenetic lineage | Measured at baseline - time of enrollment. There are no further samples or visits in the study.
  Whole genome sequencing of UK and global syphilis samples combined with phylogenomic and population genomic analyses to determine the population structure and diversity of Treponema both regionally and in global context. Diversity will be assessed by measuring nucleotide diversity between samples and reference genomes.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - University Hospitals Birmingham, Birmingham
  - Brighton and Sussex NHS Trust, Brighton
  - Leeds University Teaching Hospital, Leeds
  - Mortimer Market Centre, London
  - Penine Acute Hospitals Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided